CLINICAL TRIAL: NCT05961332
Title: COmparison of Clarus and Optos Ultrawide Field Imaging Systems for Geographic Atrophy (COCO-GA) Protocol
Brief Title: COmparison of Clarus and Optos Ultrawide Field Imaging Systems for Geographic Atrophy
Acronym: COCO-GA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2023-0958; SMPH/OPHTHAL&VIS SCI/FPRC (Other: UW Madison); Protocol Version 3/20/2025 (Other: UW Madison)
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Macular Degeneration, Age Related; Geographic Atrophy
MeSH Terms: conditions — Macular Degeneration; Geographic Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Fundus autofluorescence (FAF) imaging (Experimental)
  Interventions: Device: Spectralis FAF imaging; Device: Optos imaging; Device: Zeiss Clarus 700 imaging

INTERVENTIONS:
Device: Spectralis FAF imaging — Spectralis is a scanning laser ophthalmoscope which uses a blue light excitation wavelength of 488nm and a 500nm barrier filter to produce FAF images. Spectralis images 20-55 degrees of the retina.
Device: Optos imaging — Optos is an ultrawide field imaging platform which images up to 200 degrees of the retina. It uses both a green-light excitation wavelength of 532nm and a red-light excitation wavelength of 633nm with an emission filter of greater than 540nm to produce FAF images.
Device: Zeiss Clarus 700 imaging — Zeiss Clarus 700 is an ultrawide field imaging system with similar retinal coverage to that of Optos. It uses Broad Line Fundus Imaging to produce blue FAF images at excitation wavelengths of 435-500nm and green FAF images at wavelengths of 500-585nm

SUMMARY:
The goal of this clinical trial is to compare measurements of geographic atrophy (GA) area between several types of imaging, in order to assess accuracy. The main question to answer is which imaging device provides measurements that are most similar to the standard of care device.

Participants will be patients of a retina doctor at University Station Eye Clinic with geographic atrophy, and can expect to be in the study for 60-75 minutes.

DETAILED DESCRIPTION:
This study is a single site pilot comparative imaging study in which enrolled participants will undergo dilated fundus exam as per standard of care. Study images will be obtained using Optos ultrawide field fundus autofluorescence (FAF) and both blue and green ultrawide field FAF with Zeiss Clarus. Autofluorescence (AF) imaging will also be performed on the Spectralis as it is currently the gold standard. The goal will be to obtain all images in 60-75 minutes over one visit. Images will be assessed, and area of geographic atrophy measured independently by two experienced readers.

ELIGIBILITY:
Inclusion Criteria:

* 50 years or older and may be either male or female and may be of any race
* Established diagnosis of GA due to AMD
* GA characteristics: GA area of between 1.25 mm² and 23 mm², with seventy percent of eyes having GA area ranging from 2.5 mm² to 17.5 mm². GA may be unifocal or multifocal. GA may be subfoveal or extrafoveal, with twenty-five percent of eyes having subfoveal GA. The presence of concurrent peripapillary atrophy will not exclude subjects from participation
* Willing to participate as evidenced by signing the written informed consent

Exclusion Criteria:

* Unable to tolerate opthalmic imaging
* Presence of neovascular AMD on OCT as confirmed by an ophthalmologist
* Presence of significant media opacity preventing adequate retinal imaging
* Presence of concurrent retinal disease which may confound assessment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-10-06 (Actual); Primary Completion 2025-05-27 (Actual); Study Completion 2025-05-27 (Actual)

PRIMARY OUTCOMES:
Comparison of geographic atrophy area measurements by Clarus with standard Spectralis imaging | Up to 75 minutes
  Graders will independently measure area of GA from images of each device. The measurements (in mm²) will be compared between the two devices.
Comparison of geographic atrophy area measurements by Optos with standard Spectralis imaging | Up to 75 minutes
  Graders will independently measure area of GA from images of each device. The measurements (in mm²) will be compared between the two devices.
Comparison of geographic atrophy area measurements between Clarus and Optos | Up to 75 minutes
  Graders will independently measure area of GA from images of each device. The measurements (in mm²) will be compared between the two devices.

SECONDARY OUTCOMES:
Prevalence of atrophy outside the standard 30 degrees in Clarus and Optos ultrawide field images | Up to 75 minutes
  The presence of atrophy outside field 2 will be documented from the two ultrawide field imaging devices
Prevalence of other autofluorescence abnormalities outside the standard 30 degrees in Clarus and Optos ultrawide field images | Up to 75 minutes
  The presence of abnormal autofluorescence outside field 2 will be documented from the two ultrawide field imaging devices

CONTACTS AND LOCATIONS:
Overall Officials: Amitha Domalpally, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No